CLINICAL TRIAL: NCT04341857
Title: Phase II Clinical Study of PD-1 Monoclonal Antibody (Sintilimab) Combined With FLOT Regimen for Neoadjuvant Therapy of Gastric Adenocarcinoma/ Esophagogastric Junction Adenocarcinoma
Brief Title: PD-1 Monoclonal Antibody Combined With FLOT Regimen for Neoadjuvant Therapy of Gastric Adenocarcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HN20190929
Record Dates: First submitted 2020-04-01; First posted 2020-04-10 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Gastric and Esophagogastric Junction Adenocarcinoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sintilimab combined with FLOT regimen (Experimental): Oxaliplatin#80mg/m2d1#iv infusion for 2 hours# Calcium leucovate#200mg/m2d1#iv infusion# Fluorouracil#2600mg/m2,intravenous drip for 24h# Docetaxel#50mg/m2,intravenous drip for 1 h# Every 14 days is one cycle# Sintilimab#200mg, d1#iv infusion Every 21 days is one cycle.
  Interventions: Drug: PD-1 Monoclonal Antibody(Sintilimab)

INTERVENTIONS:
Drug: PD-1 Monoclonal Antibody(Sintilimab) — Sintilimab combined with FLOT regimen,Docetaxel#50mg/m2d1,iv infusion for 1 hour#,Oxaliplatin#80mg/m2d1#iv infusion for 2 hours#,Calcium,leucovate#200mg/m2d1#iv infusion# ,Fluorouracil#2600mg/m2,intravenous drip for 24h# Every 14 days is one cycle# Sintilimab#200mg, d1#iv infusion Every 21 days is one cycle.

SUMMARY:
This is a prospective single arm phase II clinical study to compare the safety and efficacy of PD-1monoclonal antibody +FLOT in patients with gastric adenocarcinoma/esophagus-gastric junction adenocarcinoma.

DETAILED DESCRIPTION:
Into a set of 25 cases of the gastric carcinoma confirmed by pathology or gastroesophageal junction adenocarcinoma (cT4 and/or N + M0, Multi-Disciplinary Team thought line to perioperative treatment) patients, preoperative accept four cycle by bead a resistance + sintilimab + capecitabine plus oxaliplatin into new adjuvant chemotherapy, because PD1 antibodies distance between surgery time interval is the lack of clinical data, judging by the researchers is 4 cycles of chemotherapy combination of sintilimab .The patient was able to undergo D2 radical surgery.Pathological examination was carried out to observe the pCR and the infiltration rate of immune cells.After the operation, patients continued to receive 4 cycles of capecitabine + oxaliplatin adjuvant therapy, and the total number of chemotherapy cycles was 8 cycles.Disease-free survival time and safety of treatment were observed, and OS, ORR and quality of life of all patients were followed up.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent has been signed;
* Only patients aged 18-75 were enrolled;
* Pathologically confirmed gastric adenocarcinoma (cT4 or/and N+M0, MDT considers perioperative treatment necessary) :Bone scan should be performed if bone metastasis is suspected.If peritoneal metastasis is suspected, laparoscopy should be performed;
* No previous cytotoxic chemotherapy or targeted therapy;
* No previous local resection of the tumor;
* ECOG 1 or less;
* Tumor specimens capable of detecting PDL-1 and MSI status are available.The detection of PDL-1 and MSI will be conducted after random grouping.This test requires the patient to provide a paraffin-embedded biopsy specimen;
* Leukocyte ≥ 4×109/L, platelet ≥ 100×109/L without transfusion, absolute value of neutrophils (ANC) without granulocyte stimulation factor ≥ 1.5×109/L, and hemoglobin≥ 90 g/L;
* Bilirubin ≤ 1.5 times of the upper limit of normal value, and rice grass and rice propyl transaminase ≤ 2.5 times of the upper limit of normal value;
* Serum creatinine ≤ 1.5 times the upper limit of normal value, or GFR>45ml/min;
* Serum albumin ≥ 25g /L (2.5g /dL);
* INR or aPTT ≤1.5 times ULN;

Exclusion Criteria:

* Allergy to any experimental drug and its excipients, or a history of severe allergy, or a contraindication to the experimental drug;
* Ahistory of autoimmune diseases or active stage;
* Previous allogeneic bone marrow transplantation or organ transplantation;
* Congenital pulmonary fibrosis, drug-induced pneumonia, organized pneumonia, or ct-confirmed active pneumonia;
* HIV test positive;
* Active hepatitis b or c;
* Active tuberculosis;
* Uncontrolled cancer pain;
* Live attenuated vaccine was injected within 4 weeks before the study began, or live attenuated vaccine was expected to be injected during the trial or within 5 months after the trial;
* Previous immunotherapy, including CTLA4, anti-pd-1, or anti-pdl1 monoclonal antibody;
* CT suggested active pulmonary inflammation;
* Systemic application of glucocorticoids or immunosuppressants within 2 weeks before the start of the trial.Inhaled glucocorticoids and glucocorticoids are allowed;
* There are taboos on hormone use;
* Severe cardiovascular disease, myocardial infection or cerebrovascular accident, arrhythmia, unstable angina within 3 months before the start of the trial;
* Uncontrolled increase in blood pressure or blood sugar;
* Other malignancies prior to 5 years, with the exception of cervical carcinoma in situ, non-melanoma skin cancer, or stage I uterine cancer;
* Known central nervous system metastases;
* Peripheral neuropathy ≥ NCI CTCAE grade 2;
* Serum albumin below 2.5 g/dL;
* Uncontrolled or symptomatic hypercalcemia;
* Infections requiring antibiotics within 14 days prior to the start of the trial;
* Chronic enteritis;
* Clinically significant active gastrointestinal bleeding;
* Non-diagnostic surgery within 4 weeks before the start of the trial;
* Any other disease where there is evidence of a need to restrict the use of the experimental drug;
* Participate in other tests within 30 days before the start of the test, or plan to participate in other tests during the test;
* Receive other experimental drugs within 28 days prior to the start of the trial;
* Pregnantor lactating women, or women who plan to become pregnant within 5months after the end of treatment.Women of childbearing age should undergo a blood pregnancy test within 7 days of the start of the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2019-07-30 (Actual); Primary Completion 2022-05-30 (Estimated); Study Completion 2022-07-30 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response (pCR) rate | immediately after surgery
  Complete pathological response can be determined if no tumor lesion remains or only carcinoma in situ remains in the Complete pathological response can be determined if no tumor lesion remains or only carcinoma in situ remains in the Complete pathological response can be determined if no tumor lesion remains or only carcinoma in situ remains in the surgical specimens (see WHO solid tumor efficacy criteria

SECONDARY OUTCOMES:
Disease free survival(DFS) | From the date of first treatment dose until documented disease progression or death from any cause. whichever occur first, assessed up to 30 months
  The interval between the dates of the first dose of trial treatment until first documentation of disease progression or death, whichever occurs first. Patients with new non-breast cancer malignancy must continue to be followed for progression of the original breast cancer. For patients without progression, follow-up is censored at the date of last disease assessment without progression, unless death occurs within 12 weeks following the date last known progression-free, in which case the death will be counted as a DFS event.

CONTACTS AND LOCATIONS:
Overall Officials: Ning Li, Phd, Principal Investigator — Henan Cancer Hospital
Locations (1):
- Henan Cancer Hospital, Zhengzhou, Henan, China